CLINICAL TRIAL: NCT02057848
Title: A Prospective, Randomized Trial Testing Different Regimens of Carbohydrate Administration to Prevent Hypoglycaemia During a Standardized Bout of Moderate Physical Activity in Patients With Type 1 Diabetes
Brief Title: Carbohydrates to Prevent Hypoglycaemia During Physical Activity in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael A. Nauck (Other)
Responsible Party: Sponsor-Investigator, Michael A. Nauck, Prof. Dr. med., Diabeteszentrum Bad Lauterberg im Harz
Organization: Diabeteszentrum Bad Lauterberg im Harz (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DZBL-2014-1; 2014-000561-46 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Hypoglycaemia
Keywords: carbohydrate, hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- low amount of carbohydrates (Active Comparator): 2 x 10 g carbohydrates (muesli bars)
  Interventions: Other: low amount of carbohydrates
- high amount of carbohydrates (Active Comparator): 2 x 20 g carbohydrates (muesli bars)
  Interventions: Other: high amount of carbohydrates
- Rapid-acting carbohydrates (Other): 30 g rapidly absorbable carboh. + 20 g muesli bar
  Interventions: Other: Rapid-acting carbohydrates

INTERVENTIONS:
Other: low amount of carbohydrates — different regimens of carbohydrate administration to prevent hypoglycaemia during a standardized bout of moderate physical activity in patients with type 1 diabetes
  Arms: low amount of carbohydrates
Other: high amount of carbohydrates — different regimens of carbohydrate administration to prevent hypoglycaemia during a standardized bout of moderate physical activity in patients with type 1 diabetes
  Arms: high amount of carbohydrates
Other: Rapid-acting carbohydrates — different regimens of carbohydrate administration to prevent hypoglycaemia during a standardized bout of moderate physical activity in patients with type 1 diabetes
  Arms: Rapid-acting carbohydrates

SUMMARY:
Backgrounds/Aims: It was the aim to prospectively study the optimum regime of "preventive" carbohydrate administration for prevention of hypoglycaemic episodes during a standardized bout of physical activity.

DETAILED DESCRIPTION:
Research design and methods: 24 patients with type 1 diabetes participated in one experiment without physical activity and in three experiments with a 4 km, 60 min hike starting at 2 p.m., either administering 2 x 10 g or 2 x 20 g carbohydrates (muesli bars) before starting and at 30 min (during the hike). Plasma glucose was determined with a laboratory method and additional carbohydrates needed to treat hypoglycaemia between 2 and 8 p.m. were recorded.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes mellitus, 18-75 years, BMI 18-35 kg/m², Diabetes duration > 1 year

Exclusion Criteria:

General bad health status, Malignant diseases, Systemic glucocorticoid treatment, Coronary heart disease, Uncontrolled arterial hypertension, Acute infection diseases, Diseases of liver or kidney with significant organ malfunction, Abuse of alcohol or other drugs, Participation in another trial in the last 3 months

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof. Dr., Principal Investigator — Diabeteszentrum
Locations (1):
- Diabeteszentrum, Bad Lauterberg im Harz, Germany